CLINICAL TRIAL: NCT07385547
Title: A Phase 1 Study to Assess the Effect of Renal Impairment on the Pharmacokinetics of GL0034
Brief Title: Study to Evaluate if Exposure to Drug is Impacted in Participants With Renal Insufficiency
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTRE-25-01
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GL0034 (Experimental): Single dose of GL0034
  Interventions: Drug: GL0034

INTERVENTIONS:
Drug: GL0034 — Subcutaneous (SC) administration of a single dose of GL0034

SUMMARY:
This is an open-label, single-dose, Phase 1 clinical study designed to evaluate the effect of renal impairment on the pharmacokinetics (PK) of GL0034, a long-acting GLP-1 receptor agonist. Approximately 40 adult participants will be enrolled across four groups: normal renal function, moderate renal impairment, severe renal impairment without dialysis, and severe renal impairment with dialysis. Each participant will receive a single subcutaneous dose of GL0034. Blood samples will be collected for PK analysis. Secondary objectives include assessing safety and tolerability. The study will help determine whether renal impairment affects GL0034 exposure and inform dosing recommendations for patients with compromised renal function.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to sign a written or electronic informed consent.
2. Participant is an adult male or female, aged between 18 and 80 years of age, inclusive, at the time of screening.
3. Participant has eGFR as defined by CKD-EPI equation and converted to the unit of mL/min according to the following ranges:

   * eGFR ≥ 90 mL/min;
   * eGFR ≥ 30-59 mL/min;
   * eGFR < 30 mL/min, not on dialysis;
   * eGFR < 30 mL/min, on intermittent hemodialysis.
4. Participant has a body mass index ≥ 18 kg/m2 and ≤ 42 kg/m2 at the Screening visit.
5. Contraception requirements:

   Female participants must:

   If of reproductive age and sexually active, be willing and able to use a medically highly effective form of birth control 4 weeks prior to and for 30 days following the dose of trial medication. Examples of medically highly effective forms of birth control are:
   1. Confirmed infertility due to surgical procedure or post-menopausal (cessation of menses for at least 12 months prior to Screening).
   2. Confirmed infertility of sexual partner or partner of the same sex.
   3. Hormonal contraceptive (oral, combined, patch, vaginal ring, injectable, implant) in females.
   4. Double-barrier method (any combination of physical and chemical methods).
   5. Intrauterine device with a failure rate less than 1% per year.

      Male participants must:
   6. Agree to use, with their partners, one of the highly effective contraceptive methods, from Baseline until at least 30 days following last dose of trial drug.
   7. Refrain from donating sperm during the trial and for at least 30 days after the end of the trial.
6. Participant is willing and able to comply with the study protocol, visit schedule, and other study-related instructions and procedures.

   Participants with Renal Impairment
7. The participant must have no clinically significant change in disease status within the last 30 days before screening, as documented by the participant's recent medical history.
8. The participant must have a condition consistent with renal impairment, for at least 3 months, and associated symptoms, but otherwise be determined to be in good health in the opinion of the Investigator.
9. The participant must have blood pressure (after the participant is supine for at least 5 minutes) between 90 and 160 mmHg systolic, inclusive, and not higher than 110 mmHg diastolic. If blood pressure is out of range, up to 2 repeated assessments are permitted at Screening and check-in. Pulse should not be higher than 110 beats per minute (bpm).
10. Concomitant medications to treat underlying disease states or medical conditions related to renal impairment are allowed, however must be on a stable dose of medication and/or treatment regimen for at least 4 weeks before dosing as well as during the study.

Exclusion Criteria:

1. Participant has a screening calcitonin ≥ 50 ng/L (pg/mL).
2. Participant is on continuous renal replacement therapy or peritoneal dialysis.
3. Participant has a personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome (MENS) type 2.
4. Participant has a history of pancreatitis (acute or chronic).
5. Participant is taking medications with a narrow therapeutic index such as digoxin, warfarin, etc.
6. Participant has a history of major depressive disorder within 2 years before randomization.
7. Participant has any lifetime history of a suicidal attempt.
8. Participant has any medical condition that, in the opinion of the Investigator, can confound study assessments or safety concerns.
9. Participant has a known hypersensitivity to the study medications or excipients.
10. Participant has clinically significant abnormal values on Screening laboratory tests or other evidence of uncontrolled disease involving any system-organ (e.g., cardiovascular, pulmonary, hepatic, neurological, endocrine, GI, psychiatric, etc.) that, in the opinion of the Investigator, would put the participant at risk by participating in the study.
11. Participant has a positive urine drug screen (amphetamine, barbiturate, benzodiazepine, cocaine, opiates, tetrahydrocannabinols). A positive test is allowed in case the participant receives a prescription drug responsible for the positive test. Waived for ESRD participants with no urine output.
12. Participant had a myocardial infarction, unstable angina pectoris, or ischemic stroke within the past 6 months prior to investigational product administration.
13. Participant has a clinically significant ECG abnormality as judged by the Investigator.
14. Participant has an active malignancy.

    Note: participants with past history of malignancy may be included if:
    * Participant has a history of basal cell or in-situ squamous cell carcinoma of skin that has been adequately treated and resolved, per Investigator's judgement.
    * Participant has a history of other malignancy that have been adequately treated with no evidence of recurrence/relapse within the last 5 years, per Investigator's judgement.
15. Participant has a history of alcohol or drug abuse in the previous two years.
16. Participant has any of the following laboratory abnormalities at Screening:

    * Aspartate aminotransferase or alanine aminotransferase ≥ 3 times the upper limit of normal.
    * Serum total bilirubin ≥ 1.5 mg/dL (Note: participants with elevated total bilirubin which, as per Investigator's clinical judgement, is thought to be due to Gilbert's syndrome may be included).
    * White blood cell count < 3.0 x 103/μL.
    * International normalized ratio (INR) ≥ 1.3.
    * Hemoglobin < 11.0 g/dL in participants with normal renal function or hemoglobin < 9.0 g/dL in participants with moderate or severe renal impairment.
17. Participant has a known history of coagulopathy such that SC injection will result in excessive bleeding at the injection sites.
18. Participant has a positive serology for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C. A participant who is hepatitis C virus (HCV) antibody negative can be included in the study. A participant with positive HCV antibodies shall be tested for HCV-ribonucleic acid (RNA). If tested negative, the participant can be included in the study.
19. Participant participated in another interventional study or received another investigational drug/device/biologic within 30 days or 5 half-lives (whichever is longer) of study intervention.
20. Participant has been placed in an institution on official or judicial orders.
21. Participant is related to or dependent on the Investigator, Sponsor, or study site such that a conflict of interest may arise.
22. Participant has any condition, which, in the opinion of the Investigator, precludes participation in the study (either poses an unacceptable risk to the participant or interferes with assessment/interpretation of study outcomes).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Single dose PK exposure parameters: Maximum concentration (Cmax) | From predose through 672 hours post-dose (multiple time points)
Single dose PK exposure parameters: Area under the plasma concentration-time curve (AUC) from time zero to the time of the last quantifiable concentration (AUC0-t) | From predose through 672 hours post-dose (multiple time points)
Single dose PK exposure parameters: AUC from time zero extrapolated to infinite time (AUC0-i) | From predose through 672 hours post-dose (multiple time points)

SECONDARY OUTCOMES:
Adverse events (AEs) leading to trial discontinuation and serious adverse events (SAEs). | Week 5